CLINICAL TRIAL: NCT01255202
Title: Prospective Longitudenal Study in the Prediction of Preeclampsia/Toxemia in Twin Pregnancy
Brief Title: The Prediction of Preeclampsia/Toxemia in Twin Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Svirsky Ran, Assaf-Harofeh Medical Center
Other Study IDs: 189/09
Record Dates: First submitted 2010-12-05; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Preeclampsia/Toxemia
Keywords: preeclampsia; toxemia; twin; pregnancy; pp13; prediction; kongo red
MeSH Terms: conditions — Pre-Eclampsia; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- twin preganacies

SUMMARY:
The purpose of this study is to finout whetere uterinae artery flow , PP13 and endogolin levels in the serum and kongo red in the urine can predict preeclamsia toxemia in twin pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* a women with a vaiable twin pregnany

Exclusion Criteria:

* women with thrombophilya
* women terated with anticoagolant
* women with vascular disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with twin preganacy undergoing nuchal scan in our department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe Medical Center, Zrifin, Israel